CLINICAL TRIAL: NCT06540404
Title: Effects of Traction Mobilization Techniques on Knee Joint Position Sense and Biomechanical Properties of Knee Joint Tissues
Brief Title: Effect of Knee Mobilisation on Joint Position Sense and Tissues
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: The Jerzy Kukuczka Academy of Physical Education in Katowice (Other)
Responsible Party: Principal Investigator, Polaczek Agnieszka, Principal Investigator; Master of Science, The Jerzy Kukuczka Academy of Physical Education in Katowice
Allocation: Randomized | Model: Factorial | Masking: Double | Purpose: Basic Science
Other Study IDs: 3/01/2024
Record Dates: First submitted 2024-07-27; First posted 2024-08-06 (Actual); Last update posted 2025-02-21 (Actual); Status verified 2025-02

CONDITIONS: Manual Therapy; Knee
Keywords: knee; manual therapy; healthy people; MyotonPRO

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- Control group (No Intervention): Participants in this group did not undergo any therapy.
- Pulse traction group (Experimental): Participants assigned to this group underwent second degree impulse traction of the knee joint according to the Kaltenborn concept.
  Interventions: Other: Pulse traction
- Continuous traction group (Experimental): Participants assigned to this group underwent continuous traction of the knee joint in the third degree according to the Kaltenborn concept.
  Interventions: Other: Continuous traction
- Sham therapy group (Sham Comparator): The therapist did not use traction force, the knee joint was kept in a flexed position of 40 degrees.
  Interventions: Other: Sham therapy

INTERVENTIONS:
Other: Pulse traction — The subjects underwent impulse traction of the knee joint in the second degree according to the Kaltenborn concept.
  Arms: Pulse traction group
Other: Continuous traction — The subjects underwent continuous traction of the knee joint in the third degree according to the Kaltenborn concept.
  Arms: Continuous traction group
Other: Sham therapy — The therapist did not use traction force, the knee joint was kept in a flexed position of 40 degrees.
  Arms: Sham therapy group

SUMMARY:
The aim of this study is to evaluate the effects of traction mobilizations on position sense in the knee joint and on the biomechanical properties of the knee joint tissues.

ELIGIBILITY:
Inclusion Criteria:

* no lower extremity injuries within the past year,
* no pain within the past seven days and on the day of the study,
* feeling well on the day of the study,
* no intense physical exertion on the day of the study,
* no occurrence of delayed muscle pain on the day of the study and up to three days back.

Exclusion Criteria:

* chronic diseases affecting motor skills,
* lower extremity injuries occurring within a year and treated with a physiotherapist or physician,
* complaints of pain or malaise on the day of the study,
* knee pain within the last 7 days,
* the occurrence of delayed muscle pain up to three days back,
* participation in intense physical exertion on the day of the study.

Ages: 20 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 126 (Estimated)
Dates: Start 2024-09-08 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Joint position sense | Before intervention and immediately after intervention
  A passive-active test will be used to assess the joint position sense. The parameters will be measured angular position (degree of flexion) of the knee joint in the position passively set by the researcher and in the position actively recreated by the participant in both knee joints.

SECONDARY OUTCOMES:
Biomechanical properties of knee joint tissues: Frequency | Before intervention and immediately after intervention
  The values of knee joint tissue parameters will be assessed by using MyotonPro
Biomechanical properties of knee joint tissues: Stiffness | Before intervention and immediately after intervention
  The values of knee joint tissue parameters will be assessed by using MyotonPro
Biomechanical properties of knee joint tissues: Relaxation | Before intervention and immediately after intervention
  The values of knee joint tissue parameters will be assessed by using MyotonPro
Biomechanical properties of knee joint tissues: Decrement | Before intervention and immediately after intervention
  The values of knee joint tissue parameters will be assessed by using MyotonPro
Biomechanical properties of knee joint tissues: Creep | Before intervention and immediately after intervention
  The values of knee joint tissue parameters will be assessed by using MyotonPro

CONTACTS AND LOCATIONS:
Overall Officials: Agnieszka Polaczek, MSc, Principal Investigator — The Jerzy Kukuczka Academy of Physical Education, Katowice, Poland
Locations (1):
- Motion Analysis Laboratory, The Jerzy Kukuczka Academy of Physical Education, Katowice, Poland